CLINICAL TRIAL: NCT06786884
Title: A Pilot, Randomized Controlled Trial Evaluating the Effectiveness of Paraffin Wax On Burn Patient Function, Range of Motion and Scar
Brief Title: Paraffin Wax and Exercise Prospective
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medstar Health Research Institute (Other)
Responsible Party: Principal Investigator, Bonnie Carney, Research Scientist, Assistant Professor, Principal Investigator, Medstar Health Research Institute
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STUDY00007987
Record Dates: First submitted 2025-01-06; First posted 2025-01-22 (Actual); Last update posted 2025-06-13 (Actual); Status verified 2025-06

CONDITIONS: Burn; Scar; Exercise Therapy
Keywords: paraffin wax; burn scar; scar; burn; range of motion
MeSH Terms: conditions — Burns; Cicatrix

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Exercise Therapy Only (Other)
  Interventions: Device: standard of care exercise therapy
- Exercise Therapy with Paraffin Wax Treatment (Experimental)
  Interventions: Device: paraffin wax; Device: standard of care exercise therapy

INTERVENTIONS:
Device: paraffin wax — This is the treatment group that will receive exercise and paraffin wax
  Arms: Exercise Therapy with Paraffin Wax Treatment
Device: standard of care exercise therapy — This is the group that will only receive exercise therapy and no paraffin wax.

SUMMARY:
This study is being done to test if paraffin wax can be used to improve the range of motion and function for scars across joints when used in combination with scar rehabilitation therapy sessions. For those randomized to receive it, the paraffin wax will be used alongside the participants' exercise therapy treatments. Currently, treatments that are used in addition to rehabilitation therapy for increasing range of motion across joints in the burn population are limited. By getting more information about how paraffin wax may or may not work, patients in the future that have scars may be able to be helped.

DETAILED DESCRIPTION:
If the participants agree to take part in this study, the participants scars will be looked at and the investigators will select one site that will be involved in the research. The scar will be "randomized" to the paraffin wax or no paraffin wax groups. The treatment the participants get will be chosen by chance, like flipping a coin. Neither the participants nor the study doctor will choose what treatment you get. The participants will have a 50% chance of being given either paraffin wax or not.

The study will take place in an outpatient setting. The participants will not be admitted to the hospital overnight. All patients who enter the study will be required to follow-up for regular appointments with their burn department.

Before the participants begin treatment, the participants will come in for a pre-treatment visit where the investigators will collection information about the participants scars such as pictures, range of motion measurements, non-invasive probes, non-invasive imaging (Laser doppler imaging) and questionnaires. These questionnaires will be related to the symptoms, range of motion, function, and appearance of the participants' burn scars. At the pre-treatment visit, there is an also an optional blood draw where less than 2 tablespoons of blood are collected. It is estimated this visit will take less than 1 hour. The investigators will also collect information from the medical record about prior surgical and medical history.

Exercise treatments (which the participants have previously chosen to undergo in talking with the participants doctor) will occur approximately in 1-2-week intervals depending on what the Burn Center scheduling department allows. For completion of this study, the participants will undergo 4 exercise therapy sessions which may take about 8 weeks.

At each visit, the following measurements will be captured before and after each exercise session. Those assigned to the paraffin wax group will have an additional assessment collected before their exercise therapy session and after the paraffin wax has been removed. Measurements at each visit include active and passive range of motion measurements of the affected joint, non-invasive probe measurements to measure water loss and hardness of your scar and the adjacent area of normal skin, digital photography, non-invasive laser doppler imaging (LDI), surface-level skin temperature measurements using either an infrared thermometer or skin temperature strip as well as pain and itch rating scales.

When applicable, the paraffin wax will be applied to the top of the scar for 15 minutes and repeat measurements previously listed above will be collected before your standard of care rehabilitation session. These sessions conducted by the burn rehab therapist may include scar massage, exercises, and functional activity. Specific treatments will be documented.

At each study visit, photographs will be taken of the study designated scar. All photographs taken for the purpose of this study will be taken by a high-resolution study camera. Photographs will be labeled with your study ID number. All efforts will be made to minimize the amount of identifiable information such as the participants' face or tattoos in these photos.

The procedures/treatments in this study that are considered experimental/investigation are: the use of the study product (paraffin wax) to assess the effect on burn scar that crosses an extremity joint during rehabilitation exercises.

The following procedures are part of the research study and would not normally be done as part of routine care: study provided paraffin wax and control application to the scar, scar assessments, digital photography, LDI, non-invasive imaging and measurements. These procedures are part of the study and will not be charged to insurance.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Patients with burn scar that crosses an upper or lower extremity joint (shoulder, elbow, wrist, hand, hip, knee, ankle)
* Patients that have been prescribed a rehabilitation program where paraffin wax could be used as an adjunct to rehab exercise therapy

Exclusion Criteria:

* Adults unable to provide informed consent
* Injury etiology other than burn (ex: cutaneous trauma, cold injury, etc.)
* Pregnant women
* Prisoners

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-01-06 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
Range of motion | 4th exercise session, an average of 4 weeks post enrollment
  Range of motion (degrees) of the affected joint before and after paraffin wax between the paraffin and no paraffin groups

SECONDARY OUTCOMES:
Trans-epidermal water loss | 4th exercise session, an average of 4 weeks post enrollment
  Trans-epidermal water loss (TEWL)(kg/m2h) of the HTS before and after paraffin wax between the paraffin and no paraffin groups.
  Minimum: 0 Maximum: 100 Higher score is a worse outcome.
Stiffness | 4th exercise session, an average of 4 weeks post enrollment
  Scar elasticity/hardness/stiffness by durometry (N/m) of the HTS before and after paraffin wax between the paraffin and no paraffin groups.
  Minimum: 0 Maximum: 300 Higher score is a worse outcome.
Pain visual analog scale | 4th exercise session, an average of 4 weeks post enrollment
  Pain visual analog scales (score) before and after paraffin wax between the paraffin and no paraffin groups.
  Minimum: 0 Maximum: 100 Higher score is a worse outcome.
Itch visual analog scale | 4th exercise session, an average of 4 weeks post enrollment
  Itch visual analog scales (score) before and after paraffin wax between the paraffin and no paraffin groups.
  Minimum: 0 Maximum: 100 Higher score is a worse outcome.
Scar surface temperature | 4th exercise session, an average of 4 weeks post enrollment
  Scar surface temperature (degrees celsius) before and after paraffin wax by scanner between the paraffin and no paraffin groups.
  Minimum: 0 Maximum: 100 Higher score is a worse outcome.
Patient and observer scar assessment scale | 4th exercise session, an average of 4 weeks post enrollment
  Pre and Post Study Patient and observer scar assessment scale (POSAS) version 3.0 pre and post paraffin at the first session and session four between the paraffin and no paraffin groups.
  Minimum: 0 Maximum: 10 Higher score is a worse outcome.
Perfusion | 4th exercise session, an average of 4 weeks post enrollment
  •Laser doppler imaging of perfusion (perfusion units) before and after paraffin wax first session only between the paraffin and no paraffin groups.
  Minimum: 0 Maximum: 500 Higher score is a worse outcome.
Lower extremities functional scale | 4th exercise session, an average of 4 weeks post enrollment
  • Pre (session 1) and Post (final session) study Lower extremity functional scale (LEFS) (score) between the paraffin and no paraffin groups.
  Minimum: 0 Maximum: 80 Lower score is a worse outcome.
Disabilities of the shoulder and hand | 4th exercise session, an average of 4 weeks post enrollment
  • Pre (session 1) and Post (final session) study disabilities of the arm, shoulder, and hand (DASH) (score) between the paraffin and no paraffin groups.
  Minimum: 30 Maximum: 150 Higher score is a worse outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- MedStar Washington Hosptial Center, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: No